CLINICAL TRIAL: NCT01236781
Title: Comparison of Full-Field Digital Mammography With Digital Breast Tomosynthesis Image Acquisition in Relation to Screening Call-Back Rate
Brief Title: Comparison of Full-Field Digital Mammography With Digital Breast Tomography for Screening Call-Back Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Radiology (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ACRIN PA 4006
Record Dates: First submitted 2010-11-05; First posted 2010-11-09 (Estimated); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; screening; diagnostics; diagnosis; high-risk; breast neoplasms; digital mammography; mammography; tomosynthesis; dense breasts; radiation dose; comparison; Hologic; Pennsylvania; Philadelphia; breast study; mammo; tomo; mammary
MeSH Terms: conditions — Breast Neoplasms; Disease | interventions — Vertical Dimension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: Screening (Experimental): Group A comprises 500 asymptomatic women with no history of breast cancer who are scheduled for routine screening of the breasts with FFDM.
  Interventions: Device: Screening Tomosynthesis
- Group B: Diagnostic Enriched Population (Experimental): Approximately 50 asymptomatic women with no history of breast cancer who have been informed of positive (abnormal) findings from a recent (within 30 days) FFDM screening will be recruited to Group B prior to their diagnostic imaging (e.g., diagnostic FFDM and/or ultrasound and/or other).
  Interventions: Device: Diagnostic Tomosynthesis

INTERVENTIONS:
Device: Screening Tomosynthesis — Tomosynthesis imaging sets (limited tomosynthesis set and then a sequential read with the low-dose CC view added for the tomosynthesis plus set).
  Other Names: Hologic; Dimension
  Arms: Group A: Screening
Device: Diagnostic Tomosynthesis — Tomosynthesis imaging sets (limited tomosynthesis set and then a sequential read with the low-dose CC view added for the tomosynthesis plus set).
  Other Names: Hologic; Dimension
  Arms: Group B: Diagnostic Enriched Population

SUMMARY:
This multicenter trial using Hologic digital mammography units will evaluate the specificity of 2-D full field digital mammography (FFDM) versus a combination of 2-D and 3-D tomosynthesis imaging in breast cancer screening. Specificity, in this study, will be measured by the participant call-back rate by each modality. Varying combinations of 2-D mammography and tomosynthesis projections will be evaluated to optimize the screening paradigm and limit radiation exposure when tomosynthesis is incorporated. Both prospective and retrospective imaging data will be assessed.

Hypothesis: Digital breast tomography (DBT) will improve the specificity of breast cancer screening as measured by a reduction in the call-back rate while maintaining the sensitivity of cancer detection. This improved accuracy will be achieved by the optimization of the imaging sequence and number of views obtained at a capped radiation dose in the combined DBT and 2-D screening sequence.

DETAILED DESCRIPTION:
Asymptomatic women 25 years and older with no history of breast cancer will be recruited from a prospective population of patients scheduled for screening mammography (Group A). A similar population of women called back from screening for 2-D FFDM-detected abnormalities will also be recruited to provide an enriched population of true-positive and false-positive 2-D FFDM and tomosynthesis cases (Group B). Pregnant women, women unable to tolerate compression of the breast associated with mammography, women with implants, and women with breasts too large to accommodate adequate positioning of the breast for DBT are excluded from trial participation.

A total of 550 participants will be recruited--500 women will enroll for collection of prospective imaging data in this trial (Group A); 50 additional participants, recalled for diagnostic assessment after positive screening findings, will be recruited for DBT imaging data collection and retrospective image analysis (Group B). Participating institutions for this trial will be clinical research institutions in Pennsylvania with Hologic tomosynthesis units.

ELIGIBILITY:
Inclusion Criteria:

* Women 25 years of age or older;
* No history of breast cancer;
* Group A only: Asymptomatic and scheduled for screening mammography;
* Group B only: Asymptomatic and recalled for diagnostic testing due to positive findings on recent screening using FFDM, completed within 30 days prior to registration (BI-RADS 0: additional imaging needed);
* Willing to provide a written informed consent.

Exclusion Criteria:

* Pregnancy or intent to become pregnant;
* Unable or unwilling to tolerate compression associated with mammography;
* Breast implants;
* Breasts too large to allow for adequate positioning for the DBT examination;
* Group B only: Patients with FFDM taken at screening who are unwilling or unable to submit images to ACRIN;
* Group B only: Unwilling to undergo tomosynthesis on both breasts as well as potentially additional diagnostic imaging based on tomosynthesis findings;
* Unable or unwilling to complete screening and (as necessary) diagnostic imaging at same facility;
* Tomosynthesis or mammography within 11 months prior to registration (excluding the screening mammography required for Group B).

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2011-01-04 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2013-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily F. Conant, MD, Study Chair — Hospital of University of Pennsylvania
Locations (2):
- United States (2):
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Albery Einstein Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Ray S, Chen L, Keller BM, Chen J, Conant EF, Kontos D. Association between Breast Parenchymal Complexity and False-Positive Recall From Digital Mammography Versus Breast Tomosynthesis: Preliminary Investigation in the ACRIN PA 4006 Trial. Acad Radiol. 2016 Aug;23(8):977-86. doi: 10.1016/j.acra.2016.02.019. Epub 2016 May 25. PMID 27236612
- [Result] Chen L, Ray S, Keller BM, Pertuz S, McDonald ES, Conant EF, Kontos D. The Impact of Acquisition Dose on Quantitative Breast Density Estimation with Digital Mammography: Results from ACRIN PA 4006. Radiology. 2016 Sep;280(3):693-700. doi: 10.1148/radiol.2016151749. Epub 2016 Mar 22. PMID 27002418

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Asymptomatic women 25 years and older were accrued between 1/4/2011 and 1/10/2012 at Albert Einstein Med Ctr & U Pennsylvania School of Med. 2-D FFDM and tomosynthesis images were acquired using Hologic digital mammography units. (Group A). An additional set of Women called back from screening for 2-D FFDM-detected abnormalities were recruited for an enriched population (Group B) [up to 50]
Pre-assignment Details: Study will over-accrue until 550 eligible cases are available
Groups:
- Asymptomatic Women (Screening): Asymptomatic women with no history of breast cancer who are scheduled for routine screening of the breasts with FFDM.
  Screening Tomosynthesis: Tomosynthesis imaging sets (limited tomosynthesis set and then a sequential read with the low-dose CC view added for the tomosynthesis plus set).
- Enriched Diagnostic DBT Followup (Group B): Asymptomatic women with no history of breast cancer who have been informed of positive (abnormal) findings from a recent (within 30 days) FFDM screening will be recruited to Group B prior to their diagnostic imaging (e.g., diagnostic FFDM and/or ultrasound and/or other). Group B participants will consent to DBT of both breasts as part of their diagnostic imaging work up; all screening and diagnostic images will be collected for study-related analysis.
Period: Overall Study
Arm/Group | Asymptomatic Women (Screening) | Enriched Diagnostic DBT Followup (Group B)
Started | 508 | 50
Completed | 501 | 49
Not Completed | 7 | 1
Not completed — Ineligible | 2 | 1
Not completed — Did not complete study imaging | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: Screening: Asymptomatic women with no history of breast cancer who are scheduled for routine screening of the breasts with FFDM.
  Screening Tomosynthesis: Tomosynthesis imaging sets (limited tomosynthesis set and then a sequential read with the low-dose CC view added for the tomosynthesis plus set).
- Group B: Diagnostic Enriched Population: Asymptomatic women with no history of breast cancer who have been informed of positive (abnormal) findings from a recent (within 30 days) FFDM screening will be recruited to Group B prior to their diagnostic imaging (e.g., diagnostic FFDM and/or ultrasound and/or other).
  Diagnostic Tomosynthesis: Tomosynthesis imaging sets (limited tomosynthesis set and then a sequential read with the low-dose CC view added for the tomosynthesis plus set).
- Total: Total of all reporting groups
Arm/Group | Group A: Screening | Group B: Diagnostic Enriched Population | Total
Number analyzed (Participants) | 508 | 50 | 558
Age, Continuous [Mean (Full Range); unit: years] | 55 [25 to 91] | 53 [38 to 88] | 55 [25 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 508 | 50 | 558
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 0 | 9
  Not Hispanic or Latino | 497 | 50 | 547
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 220 | 31 | 251
  White | 277 | 19 | 296
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Recall Rate in Group A Participants
Description: Each participant will undergo both FFDM and DBT examinations. Each of the two exams will be interpreted separately by readers at the participating sites and any positive finding for diagnostic followup will be considered a recall.
Time Frame: at the first imaging session
Measure: Count of Participants; unit: Participants
Groups:
- FFDM Read (Group A): Full-Field Digital Mammography (FFDM) images were read locally by a reader blinded to the results of the Digital Breast Tomography (DBT) results
- DBT Read (Group A): Digital Breast Tomography (DBT) images were read locally by a reader blinded to the results of the Full-Field Digital Mammography (FFDM) results
Arm/Group | FFDM Read (Group A) | DBT Read (Group A)
Number analyzed (Participants) | 501 | 501
Participants
  Recall for additional diagnostic imaging | 29 | 34
  Routine follow-up | 472 | 467
Statistical Analysis 1: Comparison: FFDM Read (Group A) vs DBT Read (Group A); To account for the paired nature of the design, McNemar's test will be used to compare the call-back rates. H0: assumes no difference between the tests (modalities); Test type: Equivalence — no margin is assumed; p = 0.46, McNemar — 1 degree of freedom;; Exact test

2. Secondary Outcome: Accuracy Based on Pathology Results
Description: Malignant pathologic results will be used to determine Accuracy (True Positive[Sensitivity], True Negative [Specificity], Positive and Negative Predictive values[PPV,NPV]) of FFDM and limited DBT set (digital breast two-view tomosynthesis with low-dose MLO) [Groups A and B].
  A Positive screening read had an overall site recommendation of additional Workup A Positive diagnostic read is defined as either Breast having a BIRADs score of 4 or 5 on the diagnostic read (where high BIRADS indicates higher confidence of malignancy)
Time Frame: at the first imaging session, at the Diagnostic workup (within 30 Days after Screening), and 1 year (pathologic outcome)
Population: Malignant and non-malignant are reported in separate rows for the patients so that all accuracy measures can be determined (True Positive[Sensitivity], True Negative [Specificity], Positive and Negative Predictive values[PPV,NPV])
Measure: Count of Participants; unit: Participants
Groups:
- FFDM Screening Read (Group A): Full-Field Digital Mammography (FFDM) images were read locally by a reader blinded to the results of the Digital Breast Tomography (DBT) results.
  Screening Read Positive = Recall for additional imaging
- Limited DBT Set (Digital Breast Two-view Tomosynthesis With Low-dose MLO) (Group A): Digital Breast Tomography (DBT) images were read locally by a reader blinded to the results of the Full-Field Digital Mammography (FFDM) results DBT reads used limited DBT set (digital breast two-view tomosynthesis with low-dose MLO) Screening Read Positive = Recall for additional imaging
- Full-Field Digital Mammography (FFDM) Screening Read (Group B): FFDM Screening Read results for Asymptomatic women with no history of breast cancer who have been informed of positive (abnormal) findings from a recent (within 30 days) FFDM screening will be recruited to Group B prior to their diagnostic imaging (e.g., diagnostic FFDM and/or ultrasound and/or other). Group B participants will consent to DBT of both breasts as part of their diagnostic imaging work up; all screening and diagnostic images will be collected for study-related analysis.
  Screening Read Positive = Recall for additional imaging
- DBT Diagnostic Read (Group B): DBT Diagnostic results for Asymptomatic women with no history of breast cancer who have been informed of positive (abnormal) findings from a recent (within 30 days) FFDM screening will be recruited to Group B prior to their diagnostic imaging (e.g., diagnostic FFDM and/or ultrasound and/or other). Group B participants will consent to DBT of both breasts as part of their diagnostic imaging work up; all screening and diagnostic images will be collected for study-related analysis.
  Diagnostic Read Positive =BIRADS 4 or 5
Arm/Group | FFDM Screening Read (Group A) | Limited DBT Set (Digital Breast Two-view Tomosynthesis With Low-dose MLO) (Group A) | Full-Field Digital Mammography (FFDM) Screening Read (Group B) | DBT Diagnostic Read (Group B)
Number analyzed (Participants) | 501 | 501 | 49 | 49
Participants
  Malignant (pathology): number analyzed (Participants) | 4 | 4 | 4 | 4
  Malignant (pathology): Read Positive | 3 | 3 | 4 | 4
  Malignant (pathology): Read Negative | 1 | 1 | 0 | 0
  Malignant (pathology): No exam | 0 | 0 | 0 | 0
  Not-Malignant (pathology): number analyzed (Participants) | 497 | 497 | 45 | 45
  Not-Malignant (pathology): Read Positive | 26 | 31 | 44 | 18
  Not-Malignant (pathology): Read Negative | 471 | 466 | 1 | 26
  Not-Malignant (pathology): No exam | 0 | 0 | 0 | 1

3. Secondary Outcome: Accuracy, Based on Pathology Results, by Lesion Classification
Description: Malignancy determined by pathology and follow-up will be used to determine Accuracy (True Positive[Sensitivity], True Negative [Specificity], Positive and Negative Predictive values[PPV,NPV]) of FFDM and limited DBT set (digital breast two-view tomosynthesis with low-dose MLO) with results reported by lesion-type characterization (calcification-only lesions versus soft-tissue lesions,)[Groups A and B].
  A Positive screening read had an overall site recommendation of additional screening A Positive diagnostic read is defined as either Breast having a BIRADs score of 4 or 5 on the diagnostic read.
Time Frame: as for outcome 2
Population: Malignant and non-malignant (by Pathology) are reported in separate rows for the patients so that all accuracy measures can be determined (True Positive[Sensitivity], True Negative [Specificity], Positive and Negative Predictive values[PPV,NPV])
Measure: Count of Participants; unit: Participants
Arm/Group | FFDM Screening Read (Group A) | Limited DBT Set (Digital Breast Two-view Tomosynthesis With Low-dose MLO) (Group A) | Full-Field Digital Mammography (FFDM) Screening Read (Group B) | DBT Diagnostic Read (Group B)
Number analyzed (Participants) | 501 | 501 | 49 | 49
Participants
  Non-malignant: number analyzed (Participants) | 497 | 497 | 45 | 45
  Non-malignant: Recalled calcification-only | 5 | 4 | 14 | 8
  Non-malignant: Recalled not calcification-only | 19 | 27 | 30 | 10
  Non-malignant: Not-Recalled calcification-only | 2 | 0 | 0 | 6
  Non-malignant: Not-Recalled not calcification-only | 1 | 2 | 0 | 20
  Non-malignant: No Lesions seen with modality | 470 | 464 | 1 | 1
  Malignant: number analyzed (Participants) | 4 | 4 | 4 | 4
  Malignant: Recalled calcification-only | 1 | 1 | 3 | 3
  Malignant: Recalled not calcification-only | 2 | 2 | 1 | 1
  Malignant: Not-Recalled calcification-only | 0 | 0 | 0 | 0
  Malignant: Not-Recalled not calcification-only | 0 | 0 | 0 | 0
  Malignant: No Lesions seen with modality | 1 | 1 | 0 | 0

4. Secondary Outcome: Callback Rate of Two-view Limited Tomosynthesis Set (With Low-dose MLO View Alone) With the Tomosynthesis Plus Set (Low-dose MLO View Plus Addition of Low-dose CC View)
Description: Sequential interpretation results for call- back from two-view limited tomosynthesis set (with low-dose MLO view alone) and tomosynthesis plus set (low-dose MLO view plus addition of low-dose CC view)
Time Frame: At the Diagnostic workup (within 30 Days After Screening) and up to 18-months post-screening (Pathology Measure)
Measure: Count of Participants; unit: Participants
Groups:
- Two-view Limited Tomosynthesis Set (With Low-dose MLO View Alone): Group A; Two-view Limited Tomosynthesis Set (With Low-dose MLO View Alone): Group B: Sequential interpretation results for two-view limited tomosynthesis set (with low-dose MLO view alone)
- Tomosynthesis Plus Set (Low-dose MLO View Plus Addition of Low-dose CC View): Group A; Tomosynthesis Plus Set (Low-dose MLO View Plus Addition of Low-dose CC View): Group B: Sequential interpretation results for Tomosynthesis plus set (low-dose MLO view plus addition of low-dose CC view)
Arm/Group | Two-view Limited Tomosynthesis Set (With Low-dose MLO View Alone): Group A | Tomosynthesis Plus Set (Low-dose MLO View Plus Addition of Low-dose CC View): Group A | Two-view Limited Tomosynthesis Set (With Low-dose MLO View Alone): Group B | Tomosynthesis Plus Set (Low-dose MLO View Plus Addition of Low-dose CC View): Group B
Number analyzed (Participants) | 501 | 501 | 49 | 49
Participants
  Recall for additional diagnostic imaging | 34 | 30 | 29 | 30
  Routine follow-up | 467 | 471 | 20 | 19
Statistical Analysis 1: Comparison: Two-view Limited Tomosynthesis Set (With Low-dose MLO View Alone): Group A vs Tomosynthesis Plus Set (Low-dose MLO View Plus Addition of Low-dose CC View): Group A; H0: no difference between the 2 modalities; Test type: Equivalence — no equivalence margin; p = 0.2188, McNemar — Due to the paired nature of the data an exact McNemar's Test is used; Exact test

5. Secondary Outcome: Radiation Dose
Description: Radiation dose by modality (FFDM & DBT2D/3D) Dose obtained from the data contained in the acquisition DICOM headers.
Time Frame: at the first imaging session
Measure: Mean (Standard Deviation); unit: mGy
Units Other Than Participants: views
Groups:
- FFDM Views (Group A): Full-Field Digital Mammography (FFDM) views
- DBT 2D Exam (Group A): Digital Breast Tomography (DBT) images 2D views
- DBT 3D Exam (Group A): Digital Breast Tomography (DBT) images 3D projection images
Arm/Group | FFDM Views (Group A) | DBT 2D Exam (Group A) | DBT 3D Exam (Group A)
Number analyzed (Participants) | 495 | 495 | 495
Number analyzed (views) | 2262 | 1980 | 1980
mGy | 1.79 (065) | 1.39 (0.53) | 1.84 (0.55)

6. Secondary Outcome: Regression Model Parameters for Factors Effecting Radiation Dose
Description: a mixed Regression Model to identify the determinants of participant radiation dose, including covariates (X) such as: kVp, mAs, target/filter combination, and breast thickness and compression.
  Dose = B1*X1 + B2*X2 + B3*X3 + ...
  The outcome measures is are the estimated coefficients (B) of the covariate (X) in the mixed regression model.
  The coefficient (B) of the term (X) represents the change in the mean response (dose) for one unit of change in that term. If the coefficient is negative, as the term increases, the mean value of the response decreases. If the coefficient is positive, as the term increases, the mean value of the response increases.
  Note: the TUNGSTEN/SILVER categorical target/filter combination is used as the reference category and will have a parameter value of 0.
Time Frame: at the first imaging session
Population: Dose and associated parameters were pulled from each collected images DICOM header.
Measure: Mean (Standard Deviation); unit: regression slope (Betas)
Units Other Than Participants: Images
Groups:
- FFDM Images (Group A): Full-Field Digital Mammography (FFDM) images
- DBT Images: Digital Breast Tomography (DBT) images (Group A)
Arm/Group | FFDM Images (Group A) | DBT Images
Number analyzed (Participants) | 495 | 495
Number analyzed (Images) | 2262 | 3951
regression slope (Betas)
  Intercept | -3.1852 (0.1045) | -5.3837 (0.08977)
  Exposure (mAs) | 0.01215 (0.000094) | 0.009873 (0.000103)
  KVp | 0.1384 (0.005604) | 0.2180 (0.005328)
  Anode/Filter: MOLYBDENUM/MOLYBDENUM | 0.8294 (0.02557) | NA (NA) — This anode/filter combination was not used
  Anode/Filter: MOLYBDENUM/RHODIUM | 0.5881 (0.02698) | NA (NA) — This anode/filter combination was not used
  Anode/Filter: TUNGSTEN/ALUMINUM | NA (NA) — This anode/filter combination was not used | 0.3502 (0.02885)
  Anode/Filter: TUNGSTEN/RHODIUM | -0.4400 (0.01767) | -0.1986 (0.01981)
  Anode/Filter: TUNGSTEN/SILVER | 0 (0) | 0 (0)
  Compression Force (N) | 0.000691 (0.000090) | 0.000241 (0.000099)
  Breast thickness(mm) | -0.01328 (0.001096) | -0.01362 (0.001125)

7. Secondary Outcome: Identification and Characterization of Lesion(s) Using Screening Tomosynthesis (Group A)
Description: Group A, screening tomosynthesis, cases will be evaluated using 2 methodologies. Readers will read each screening exams using either (1) the limited tomosynthesis set (with low-dose MLO view alone) or (2) the tomosynthesis plus set (low-dose MLO view plus addition of low-dose CC view) and classify the lesions they are able to visualize per SOC.
  SOC Lesions characterizations include: Calcification Only lesion , Mass, Focal Asymmetry, Architectural Distortion, Global Asymmetry, Calcification) The characterizations will be tabulated by whether or not each lesion was classified in the given category.
Time Frame: At the Diagnostic workup (within 30 Days After Screening)
Population: Analysis is base on the lesions found with either viewing method. 1 finding classified as "calcifications only" in the tomosynthesis plus set was classified as a MASS in the two-view limited tomosynthesis set
  1 finding classified as "calcifications only" in the tomosynthesis plus set was classified as a ASYMMETRY the two-view limited tomosynthesis set
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Groups:
- Method 1: Two-view Limited Tomosynthesis Set (With Low-dose MLO View Alone): In Method 1, Reader will provide sequential interpretation results for two-view limited tomosynthesis set (with low-dose MLO view alone)
- Method 2: Tomosynthesis Plus Set (Low-dose MLO View Plus Addition of Low-dose CC View): In Method 2: Reader will provide sequential interpretation results for Tomosynthesis plus set (Using the low-dose MLO view plus addition of low-dose CC view)
Arm/Group | Method 1: Two-view Limited Tomosynthesis Set (With Low-dose MLO View Alone) | Method 2: Tomosynthesis Plus Set (Low-dose MLO View Plus Addition of Low-dose CC View)
Number analyzed (Participants) | 501 | 501
Number analyzed (lesions) | 75 | 75
lesions
  CALCIFICATION ONLY LESION: Yes | 20 | 22
  CALCIFICATION ONLY LESION: No | 55 | 53
  MASS: Yes | 39 | 37
  MASS: No | 36 | 38
  FOCAL ASYMMETRY: Yes | 14 | 18
  FOCAL ASYMMETRY: No | 61 | 57
  ARCHITECTURAL DISTORTION: Yes | 2 | 2
  ARCHITECTURAL DISTORTION: No | 73 | 73
  CALCIFICATIONS: Yes | 1 | 1
  CALCIFICATIONS: No | 74 | 74
  GLOBAL ASYMMETRY: Yes | 0 | 0
  GLOBAL ASYMMETRY: No | 75 | 75

ADVERSE EVENTS:
Time Frame: 30 days from screening imaging visit
Groups:
- Asymptomatic Women (Screening) - Group A: Asymptomatic women with no history of breast cancer who are scheduled for routine screening of the breasts with FFDM.
- Enriched Cohort - Group B: An additional set of Women called back from screening for 2-D FFDM-detected abnormalities were recruited for an enriched population (Group B) [up to 50] Asymptomatic women with no history of breast cancer who have been informed of positive (abnormal) findings from a recent (within 30 days) FFDM screening. Group B participants will consent to DBT of both breasts as part of their diagnostic imaging work up
Arm/Group | Asymptomatic Women (Screening) - Group A | Enriched Cohort - Group B
All-Cause Mortality (participants affected / at risk) | 0/501 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/501 | 0/49
Other Adverse Events (participants affected / at risk) | 0/501 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2010-06-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT01236781/Prot_SAP_000.pdf
  • Informed Consent Form (2010-06-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT01236781/ICF_001.pdf